CLINICAL TRIAL: NCT06876701
Title: The Treatment of Newly Diagnosed CD19+Mixed Phenotype Acute Leukemia in Adults
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-AML-KXX
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Evaluation of the efficacy and safety of the combination of injectable bevacizumab, low-intensity chemotherapy, and venula in the treatment of newly diagnosed CD19+mixed phenotype acute leukemia in adults

SUMMARY:
Evaluation the efficacy and safety of the combination of injectable bevacizumab, low-intensity chemotherapy, and venula in the treatment of newly diagnosed CD19+mixed phenotype acute leukemia in adults

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand this study, voluntarily participate and sign an informed consent form (ICF);
2. Age: 18-75 years old (including boundary values of 18 and 75);
3. Clinically diagnosed adult Mixed Phenotype Acute Leukemia (WHO 2016 criteria) patients with CD19 positivity

Exclusion Criteria:

The subject's previous history of anti-tumor treatment meets one of the following conditions:

1. Individuals who have previously received bevacizumab
2. Individuals who have received CAR-T therapy or other gene modified cell therapies prior to screening;
3. Within 5 half lives of the first use of the investigational drug, having received anti-tumor treatment including surgery, chemotherapy, targeted therapy, or participating in other clinical trials and receiving clinical trial medication;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Negative conversion rate of evaluable residual lesions (MRD) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhaxin integrated hospital of traditional Chinese and Western Medicine, Shanghai, China